CLINICAL TRIAL: NCT04291274
Title: Long Term Neurobehavioral Effects of Anesthetics and Cochlear Implantation on Infants With Hearing Impairment
Brief Title: The Neurobehavioral Effects of Anesthetics on Infants With Hearing Impairment（Retrospective Research）
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, associate chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H-2019-T293-2
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2020-02

CONDITIONS: Long Term Neurobehavioral Effects
Keywords: infant; anesthesia; neurobehavioral development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inhalation anesthesia group: Unilateral and Bilateral cochlear implantation,which used inhalation anesthesia
- intravenous anesthesia group: Unilateral and Bilateral cochlear implantation, which used intravenous anesthesia

SUMMARY:
The long-term effect of general anesthesia on developing brain is the focus of clinicians when infants exposed to general anesthesia for a long time during operation. A retrospective study showed that children exposed to long-term or repeated operations, the anesthetics had a higher incidence of cognitive impairment in adolescence than those did no. When infants with hearing impairment undergo bilateral cochlear implant surgery, they are at high risk of long-term neurobehavioral abnormalities caused by anesthesia. In this study, investigators intend to observe the long-term behavioral abnormalities of hearing-impaired infants after intravenous or inhalation anesthesia by a ambispective cohort study.

DETAILED DESCRIPTION:
Gesell development scale contains five subscales including adaptability, fine motor, gross motor, language, and social skill evaluation. Developmental quotient (DQ) = (development age/actual age)×100. Total DQ is the average of five DQ of subscales. DQ≥86 is normal, 76≤DQ≤85 is suspicious, 55≤DQ≤75 is mild neurological damage, 40≤DQ ≤54 is moderate neurological damage, 25 B DQ B 39 is severe neurological damage, and DQ< 25 is very severe neurological damage.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing cochlear implantation under general anesthesia
* 6 to 36-month-old child
* Normal body weight
* Children with normal structures of the inner ear and auditory nerve
* Children without contraindications to anesthesia and surgery
* Patients who have not participated in other clinical trials
* Without any acute infectious diseases or systematic diseases

Exclusion Criteria:

* The participants with a Gesell score (fine motor and gross motor) lower than 86 after preoperative evaluation.
* With other illness which could affects curative effect of recovery, such as inner ear malformations (except for large vestibular aqueduct syndrome), auditory vestibular nerve dysplasia, dysgnosia and mental disease;
* Inability to cooperate with the hearing evaluation and the language training
* Cute and chronic otitis media and mastoiditis, unhealed tympanic membrane perforation
* Abnormal structure of brain, including white matter dysplasia, Demyelinating Diseases

Ages: 6 Months to 36 Months | Sex: All
Age Groups: Child
Study Population: Children undergoing cochlear implantation under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
change of Baseline Gesell Developmental Scale after 6 month | change in 6 months after surgery]
  Neurobehavior effects was measured use Gesell Developmental Scale. DQ (Developmental quotient) was calculated by (development age/actual age)×100. Total DQ is the average of five DQ of subscales. DQ≥86 is normal, 76≤DQ≤85 is suspicious, 55≤DQ≤75 is mild neurological damage, 40≤DQ≤54 is moderate neurological damage, 25≤DQ≤39 is severe neurological damage, and DQ <25 is very severe neurological damage

CONTACTS AND LOCATIONS:
Overall Officials: Jingjie Li, M.D, Study Chair — Shanghai No.9 People's Hospital
Locations (2):
- China (2):
  - Shanghai ninth people's hospital, Shanghai
  - Shanghai No.9 People's Hospital, Shanghai

REFERENCES:
- [Derived] Zhang L, Cheng Y, Xue Z, Li J, Wu N, Yan J, Wang J, Wang C, Chen W, Zhou T, Qiu Z, Jiang H. Sevoflurane impairs m6A-mediated mRNA translation and leads to fine motor and cognitive deficits. Cell Biol Toxicol. 2022 Apr;38(2):347-369. doi: 10.1007/s10565-021-09601-4. Epub 2021 Apr 29. PMID 33928466